CLINICAL TRIAL: NCT02199639
Title: Multidisciplinary Evaluation of Patients With Hemophilia of Spain, El Salvador and Bolivia. An Observational Study
Brief Title: Transcultural Multidisciplinary Evaluation of Patients With Hemophili
Acronym: ibHEro
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, RUBÉN CUESTA-BARRIUSO, PhD, Universidad Católica San Antonio de Murcia
Other Study IDs: ibHEro; ibHEro
Record Dates: First submitted 2014-07-23; First posted 2014-07-24 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2014-03

CONDITIONS: Patients With Haemophilia
Keywords: Haemophilia; Arthropathy; Range of Movement; Strength; Proprioception; Gait; Quality of Life
MeSH Terms: conditions — Hemophilia A; Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Spain: Group of patients with hemophilia recruited in the Region of Murcia (Spain) and evaluated in the Universidad Católica San Antonio between June and July 2014.
- El Salvador: Group of patients with hemophilia recruited in the city of San Salvador (El Salvador) and evaluated in the Hospital Nacional Rosales and the Hospital Nacional de niños "Benjamín Bloom" from San Salvador in April 2014.
- Bolivia: Group of patients with hemophilia recruited in the city of Santa Cruz (Bolivia) and evaluated at the Hospital Nacional de niños in Santa Cruz August 2014.

SUMMARY:
Multidisciplinary evaluation of patients with hemophilia Spain, El Salvador and Bolivia. It aims to analyze and evaluate the skeletal muscle of patients affected with hemophilia Spain, El Salvador and Bolivia; describe deficit mobility and muscular strength, depending on the degree of injury, age, presence of inhibitors and the development of physical activity; identify the relationship between the functional deficit by clinical assessment performed with the use of validated measurement scales, the assessment of the degree of injury to specific scales of hemophilia; detect biomechanical alterations of the lower limbs and their impact on gait in patients with hemophilia; and evaluate the factors that influence the perception of illness and quality of life of patients with hemophilia.

DETAILED DESCRIPTION:
Descriptive study of joint involvement in patients with hemophilia Spain, El Salvador and Bolivia.

Descriptive study of abnormal joint mobility and muscle strength as a result of acute conditions or the development of chronic articular sequelae.

Descriptive study of biomechanical changes in lower limb joints and their impact on gait in patients with hemophilia.

Descriptive study of the overall articular involvement (crepitus, pain, biomechanical and functional changes) in patients with hemophilia.

Descriptive study of the relationship between skeletal muscle pathology in patients with hemophilia and their perception of it, and their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemophilia A and B.
* Patients of all ages (pediatric, adolescents, youth and adults).
* With or without joint involvement clinically diagnosed, and with or without a previous history of hemarthrosis joint load legs.
* Patients with or without inhibitors.

Exclusion Criteria:

* Patients without prior ambulation capacity.
* Patients diagnosed with other congenital coagulopathy (von Willebrand disease, etc..).
* Patients with neurological or cognitive impairments that prevent understanding the questionnaires and physical tests.

Ages: 6 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with haemophilia from Spain, El Salvador and Bolivia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of range of motion of elbow, knee and ankle | Screening visit
  We will use a goniometric evaluation, along the lines indicated by Querol for assessing the range of motion in patients with hemophilia
Assessment of muscle strength of arm, thigh and leg | Screening visit
  We will use a measure of muscular balance with the guidelines outlined by Daniels, with the adaptation of Querol for assessing muscle strength in patients with hemophilia
Assessment of perception of joint pain | Screening visit
  We will use the visual analogue scale (VAS) for the assessment of joint pain in patients with hemophilia, with a scale from 0 (no pain) to 10 (maximum pain).
Assessment of the status joint | Screening visit
  We will use the specific questionnaire haemophilia: Haemophilia Joint Healts Score (HJHS) for the assessment of joint status
Evaluation of the performance of activities of daily living | Screening visit
  We will use the questionnaire Haemophilia Activities List (HAL), specific for patients with hemophilia
Assessment of physical performance of patients with hemophilia | Screening visit
  We will use the Physical Functioning scale (HEP-Test-Q), specific for patients with hemophilia
Assessment of personality traits of children | Screening visit
  We will use the questionnaire Eysenck Personality Questionnaire Junior (EPQJ)
Evaluation of perceived quality of life for patients with hemophilia | Screening visit
  We will use the Hemophilia-QoL and the Child Health and Illness Profile (CHIP-CE) questionnaires for children; and the Hemophilia-QoL and A36 and 36 Health Survey (SF36) questionnairesfor adults .

SECONDARY OUTCOMES:
Clinical variables of patients with hemophilia | Screening visit
  Age (years); weight (kg); Size (cm); type of haemophilia (A or B); severity of hemophilia (severe / moderate / mild); pharmacological treatment (prophylactic / on demand); presence of inhibitors; central venous catheter; family history of hemophilia; hemarthrosis in the last month; arthropathy diagnosed in some joint; use of orthoses
Socio-demographic variables of patients with hemophilia | Screening visit
  Number of hospital visits per year (reason); Distance to hospital (km); Academic formation of the patient (university studies / vocational training / basic studies / no studies); academic formation of the parents (university studies / vocational training / basic studies / no studies); patient employment (self-employment / employment has as an employed person / unemployed / retirement); parents employment (self-employment / employment has as an employed person / unemployed / retirement);

CONTACTS AND LOCATIONS:
Overall Officials: RUBEN CUESTA-BARRIUSO, PhD, Principal Investigator — Universidad Católica San Antonio
Locations (1):
- Universidad Católica San Antonio de Murcia, Murcia, Murcia, Spain